CLINICAL TRIAL: NCT06405724
Title: Comparison of the Ultrasound-guided Paravertebral Nerve Block With Liposomal Bupivacaine Versus Ropivacaine for Post-Surgical Pain After Video-Assisted Thoracoscopic Surgery:A Single-Center, Prospective, Randomized, and Controlled Trial
Brief Title: Comparison of the Ultrasound-guided Paravertebral Nerve Block With Liposomal Bupivacaine Versus Ropivacaine for Post-Surgical Pain After Video-Assisted Thoracoscopic Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TJ-IRB202403005
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Analgesia
Keywords: paravertebral nerve block; liposomal bupivacaine; video-assisted thoracoscopic surgery
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Liposomal bupivacaine (Experimental): Experimental group will receive PVB with LB 20 mL.
  Interventions: Drug: Liposomal bupivacaine
- Drug:ropivacaine (Active Comparator): Comparator group will receive PVB with 20 mL of 0.5% ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — 133mg LB 20mL thoracic paravertebral nerve block
  Other Names: Exparel
  Arms: Drug: Liposomal bupivacaine
Drug: Ropivacaine — 0.5% ropivacaine 20mL thoracic paravertebral nerve block
  Arms: Drug:ropivacaine

SUMMARY:
Prospective, randomized, and controlled trial to compare the postoperative pain management of paravertebral nerve block with liposomal bupivacaine to ropivacaine in patients undergoing elective thoracoscopic surgery.

DETAILED DESCRIPTION:
The objective of this study is to validate the analgesic efficacy of liposomal bupivacaine (LB) compared with ropivacaine when injected for paravertebral nerve block (PVB) for video-assisted thoracoscopic surgery (VATS).

We hypothesize that LB will be superior to ropivacaine in terms of postoperative pain control following VATS. The primary outcome of this study will be NRS pain scores for resting pain and NRS pain scores for cough pain 24 hours following surgery. Secondary outcomes will include pain scores over the first 120 hours following surgery, opioid consumption, opioid-related adverse events, block-related adverse events, time of first getting out of bed, catheter indwelling time, postoperative hospitalization time, patient satisfaction, and chronic pain at 1, 3, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-64 years old
2. Elective unilateral thoracoscopic surgery
3. Hospital stay ≥3 days
4. Able to cooperate in completing interviews and scale assessments
5. American Society of Anesthesiologists (ASA) classification I-III
6. Signed informed consent form

Exclusion Criteria:

1. History of thoracic surgery within the past 6 months
2. Pre-existing history of chronic pain or acute pain in the surgical area
3. Allergy to local anesthetics
4. Contraindications to thoracic paravertebral nerve block
5. Mental disorders, intellectual disabilities, epilepsy, or other neurological conditions
6. Severe heart or lung diseases
7. History of opioid drug abuse or substance abuse
8. Postoperative intubation
9. Recent participation in other clinical studies

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
pain score at rest | 24 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 24 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").

SECONDARY OUTCOMES:
pain score at rest | 6 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 6 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score at rest | 48 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 48 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 72 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score at rest | 72 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score at rest | 96 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 96 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score at rest | 120 hours after surgery
  The pain score at rest will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
pain score during coughing | 120 hours after surgery
  The pain score during coughing will be assessed using the Numeric Rating Scale (NRS), which ranges from 0 (representing "no pain") to 10 (representing "the worst pain").
Consumption of analgesic drugs | 120 hours after surgery
  the amount of analgesic drugs will be recorded
Nerve block related adverse events | 120 hours after surgery
  Any adverse event resulting from a nerve block, such as toxicity, allergic reactions, or nerve injuries, will be considered causally related.
Block duration: first reported pain | 24 hours after surgery
  Definition: timing begins at block performance
Presence of pain 1 month after surgery assessed using the Brief Pain Inventory. | 1 month after surgery
  yes/no
Presence of pain 3 months after surgery assessed using the Brief Pain Inventory. | 3 months after surgery
  yes/no
Presence of pain 6 months after surgery assessed using the Brief Pain Inventory. | 6 months after surgery
  yes/no
Hospital Anxiety and Depression Scale, HADS | day1 before surgery
  The Hospital Anxiety and Depression Scale (HADS) is primarily used to screen for anxiety and depression in general hospital patients. The HADS includes a total of 14 items, with 7 items assessing depression and 7 items assessing anxiety. There are six reverse question entries, five on the depression subscale and one on the anxiety subscale.
Insomnia Severity Index, ISI | day1 before surgery
  The Insomnia Severity Index (ISI) is a self-assessment tool for self-perception of insomnia symptoms in the past two weeks. It includes 7 items, with each item scoring 0 to 4 points. The questions involve the subject's subjective evaluation of sleep quality, including the severity of symptoms and their satisfaction with their sleep patterns. The impact of insomnia on daily functioning, the subject's awareness of the impact of insomnia on themselves, and the level of depression caused by sleep disorders.
Charlson Comorbidity Index, CCI | day1 before surgery
  The Charlson Comorbidity Index (CCI) is a commonly used evaluation method in clinical research to assess the health status of patients and predict their life expectancy by scoring coexisting diseases and age.
Mini-cog | day1 before surgery
  The Mini-Cog uses recall and clock-drawing tests to determine whether patients have cognitive impairments. A score of 0-2 indicates a positive dementia screening, while a score of 3-5 implies a negative screening, necessitating further evaluation.
Complications within 120hours after surgery | Five days after surgery
  Complications will be recorded.
The douleur neuropathique 4 questionnaire(DN4) | day1 before surgery
  This questionnaire serves as a diagnostic tool for identifying neuropathic pain. It comprises 10 options, consisting of 7 self-assessment items that evaluate symptoms. The total score is 10 points, and a score of ≥ 4 indicates the possibility of neuropathic pain, while a score < 4 rules out neuropathic pain.
The douleur neuropathique 4 questionnaire(DN4) | 1 month after surgery
  This questionnaire serves as a diagnostic tool for identifying neuropathic pain. It comprises 10 options, consisting of 7 self-assessment items that evaluate symptoms. The total score is 10 points, and a score of ≥ 4 indicates the possibility of neuropathic pain, while a score < 4 rules out neuropathic pain.
The douleur neuropathique 4 questionnaire(DN4) | 3 months after surgery
  This questionnaire serves as a diagnostic tool for identifying neuropathic pain. It comprises 10 options, consisting of 7 self-assessment items that evaluate symptoms. The total score is 10 points, and a score of ≥ 4 indicates the possibility of neuropathic pain, while a score < 4 rules out neuropathic pain.
The douleur neuropathique 4 questionnaire(DN4) | 6 months after surgery
  This questionnaire serves as a diagnostic tool for identifying neuropathic pain. It comprises 10 options, consisting of 7 self-assessment items that evaluate symptoms. The total score is 10 points, and a score of ≥ 4 indicates the possibility of neuropathic pain, while a score < 4 rules out neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China